CLINICAL TRIAL: NCT06627699
Title: Prospective, In-Vivo, Post-Market Safety and Efficacy Surveillance Registry of the MAXX Orthopedics, Freedom Total Knee® System
Status: Not yet recruiting | Type: Observational
Sponsor: Maxx Orthopedics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PK-00002
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthristis; Total Knee Anthroplasty
Keywords: Registry; Primary TKA; Total Knee Arthroplasty; Total Knee Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving the Maxx Freedom Total Knee System for primary TKA: TARGETED PATIENTS Adult male and female patients greater than 18 years of age Candidate for primary TKA GENERAL EXCLUSIONS Active infection Revision / conversion TKA (Prior UKA or HTO)
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — Post-Market Surveillance of the Freedom Total Knee System for Primary TKA

SUMMARY:
In an effort to satisfy regulatory requirements for post-market surveillance of product safety and efficacy, a representative sample of patients will be recruited for prospective monitoring.

DETAILED DESCRIPTION:
In an effort to satisfy regulatory requirements for post-market surveillance of product safety and efficacy, a representative sample of patients will be recruited for prospective monitoring.

To maintain equal site distribution per device, patient recruitment will include up to a total of twenty (20) registry sites and thirty (30) primary TKA candidates per site / surgeon for a total of 600 registry patients. A total of no more than 200 patients across all sites will be recruited per level of constraint (e.g.: 200 CR, 200:PS, 200:UC) for this registry with a 10-month accrual target from study initiation per site (~3 patients consented / month).

ELIGIBILITY:
INCLUSION CRITERIA:

Candidates for this registry must meet ALL of the following criteria:

* Patient is > 18 years of age
* Patient has failed attempts at non-operative conservative therapy
* Patient has participated in the informed consent process and signed an IRB approved informed consent
* Patient is scheduled to undergo unilateral or bilateral primary TKA of the knee

EXCLUSION CRITERIA:

Candidates will be excluded from the evaluation if ANY of the following apply:

* Patients with previous TKA, UKA, HTO or knee fusion of the indicated knee
* Patients that have undergone previous surgery of indicated knee for tumor, trauma or fracture
* Evidence of active or suspected (systemic or local) infection at time of surgery
* Other significant disabling problems from the musculoskeletal system than in the knee (i.e.: muscular dystrophy, polio, neuropathic joints)
* Patients with or having; malignancy - active malignancy, Paget's disease, renal osteodystrophy, immunologically suppressed, sickle cell anemia and systemic lupus erythematosus
* Patients with neuromuscular or neurosensory deficit
* Women who are pregnant
* Prisoner or transient
* Recent history of known narcotic abuse
* Any significant psychological disturbance past or present, that could impair the consent process or ability to complete subject self-report questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population will consist of adult male and female subjects who are suffering from moderate to severe symptoms of the following diagnoses: painful degenerative knee disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Device Survivorship | 2 years
  Revision / re-operation post-operatively due to device / device composite failure. An anticipated benefit of the device is that it is more conforming at higher degrees of flexion, which could potentially result in reduced polyethylene wear and improved survivorship over the longer-term. To assess this aspect of the device in addition to safety over the short-, intermediate- and long-term, survivorship analyses will be conducted at the targeted follow-up landmark timepoints.
  There will be 3 survivorship endpoints:
  * Revision of any component (including insert) for any reason
  * Revision of any component (including insert) for any reason except infection

SECONDARY OUTCOMES:
Original Knee Society Scale (KSS) | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  The Knee Society Score rating system was first introduced during the late 1980's and has become the standard clinical evaluation system for reporting results for patients undergoing Total Knee Arthroplasty. Most major journals strongly encourage that total knee manuscripts include Knee Society Score rating scores as part of the result section. The Knee Society Score consists of points given for pain, range of motion, and stability. The Function Score consists of points given for the ability to walk on level surfaces, and the ability to ascend and descend stairs, with deductions for the use of external supporting devices.
Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS-JR) | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  The KOOS-JR is self-administered and assesses three domains: stiffness (1 question), pain (4 questions), function / daily living (2 questions). The KOOS-JR meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome. Each item (questions) is coded from 0 to 4. The raw responses are summed (0-28) which is then converted to an interval score based on the KOOS-JR conversion table. The score is a percentage score from 0 to 100, 0 representing total knee disability and 100 representing perfect knee health.
Patient Reported Outcomes Measurement Information System (PROMIS Global-10) | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  The Patient Reported Outcomes Measurement Information System (PROMIS Global-10) is a valid and reliable patient assessment and consists of ten (10) items that measure physical health, physical functioning, general mental health, emotional distress, satisfaction with social activities and relationships, ability to carry out usual social activities and roles, pain, fatigue and overall quality of life. The response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient. The PROMIS 10 scores are predictive of healthcare utilization, mortality in general and disease-specific clinical populations.
Visual Analog Scale (VAS) | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  This scale has been designed to give subjective pain information as to the degree of knee pain you the patient is currently experiencing. VAS scoring is included in the PROMIS GLOBAL-10 assessment and is not necessary to collect a separate assessment. Applying the VAS, the patient will select a number from 1 (no pain) to 10 (maximum pain) that most closely describes their current pain.
Forgotten Joint Score (FJS-12) | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  The 12 question Forgotten Joint Score (FJS-12) was introduced with the aim of assessing the patients 'joint awareness'. The authors of the score suggest the "higher the score" is more representative of higher-level function after surgery, as to be able to forget about the joint requires the absence of pain and the ability to perform all desired functional tasks without limitation.

OTHER OUTCOMES:
Radiography (plain-film radiography as per standard of care - independent collective site assessment) | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  * Evidence of correct component position
  * Evidence of stable component fixation
  * Review of incidence and location of any lucencies, sclerotic lines, component subsidence and/or osteolysis
Adverse Events | 3-6 Weeks, 3 Months, 6 Months, 12 Months, 24 Months
  * Local (wound and skin)
  * Systemic (infection markers)
  * Clinical / radiographic evidence of component / composite failure
  * Unscheduled re-visit or re-operation within 24 months post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Asit Shah, MD, PhD, Study Chair — Chief of Orthopedics, Englewood Hospital
Locations (2):
- United States (2):
  - Ascentist Healthcare, Leawood, Kansas
  - South Texas Bone & Joint Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Proprietary nature of data for use for FDA De-Novo Submission following study conclusion.

REFERENCES:
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Thomsen MG, Latifi R, Kallemose T, Barfod KW, Husted H, Troelsen A. Good validity and reliability of the forgotten joint score in evaluating the outcome of total knee arthroplasty. Acta Orthop. 2016 Jun;87(3):280-5. doi: 10.3109/17453674.2016.1156934. Epub 2016 Mar 3. PMID 26937689
- [Background] Shim J, Hamilton DF. Comparative responsiveness of the PROMIS-10 Global Health and EQ-5D questionnaires in patients undergoing total knee arthroplasty. Bone Joint J. 2019 Jul;101-B(7):832-837. doi: 10.1302/0301-620X.101B7.BJJ-2018-1543.R1. PMID 31256677
- [Background] Lyman S, Lee YY, Franklin PD, Li W, Cross MB, Padgett DE. Validation of the KOOS, JR: A Short-form Knee Arthroplasty Outcomes Survey. Clin Orthop Relat Res. 2016 Jun;474(6):1461-71. doi: 10.1007/s11999-016-4719-1. Epub 2016 Feb 29. PMID 26926773
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- See also: Registry sponsor home page — https://maxxortho.com